CLINICAL TRIAL: NCT01037491
Title: Comparison of Ulcer Healing in Patients Taking Rabeprazole Plus Aspirin Versus Rabeprazole Plus Clopidogrel for Acute Peptic Ulcer
Brief Title: Comparison of Ulcer Healing in Patients Taking Rabeprazole With Different Antiplatelets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Fang-Yue Lin, Superintendent, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGH97-10-04
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Gastric Ulcer; Duodenal Ulcer
Keywords: aspirin, clopidogrel, peptic ulcer, proton pump inhibitor, rabeprazole, ulcer bleeding
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Peptic Ulcer | interventions — Rabeprazole; Clopidogrel

ARMS (2):
- aspirin (Active Comparator): Patients who have taken aspirin for more than 1 month and are found to have PUD by upper endoscopy will receive PPI (rabeprazole 20 mg once daily) to treat their PUD.patients will be randomly assigned rabeprazole (20 mg/day) plus aspirin (100 mg/day) or rabeprazole (20 mg/day) plus clopidogrel (75 mg/day) for 12 weeks.
  Interventions: Drug: rabeprazole plus aspirin versus rabeprazole plus clopidogrel
- clopidogrel (Active Comparator): Patients who have taken aspirin for more than 1 month and are found to have PUD by upper endoscopy will receive PPI (rabeprazole 20 mg once daily) to treat their PUD.patients will be randomly assigned rabeprazole (20 mg/day) plus aspirin (100 mg/day) or rabeprazole (20 mg/day) plus clopidogrel (75 mg/day) for 12 weeks.
  Interventions: Drug: rabeprazole plus aspirin versus rabeprazole plus clopidogrel

INTERVENTIONS:
Drug: rabeprazole plus aspirin versus rabeprazole plus clopidogrel — The primary end point is treatment success (ulcer healing rate). The secondary end point is incidence of ulcer bleeding within 12 weeks.

SUMMARY:
Clopidogrel causes significantly less peptic ulcer disease (PUD) and ulcer bleeding than low-dose aspirin in general population. However, clopidogrel is not safe enough for gastrointestinal (GI) mucosa in patients who had past history of aspirin-associated ulcer or ulcer bleeding. Aspirin plus proton pump inhibitor (PPI) is superior to clopidogrel alone in preventing recurrent ulcer bleeding in these high risk patients.

This study is to compare the ulcer healing rate and ulcer bleeding at 12 weeks in patients with aspirin-associated PUD when they take PPI (rabeprazole 20 mg/day) to treat their PUD and simultaneously take aspirin or clopidogrel for their cardiovascular (CV) prevention. Two hundred patients will be randomly assigned rabeprazole (20 mg/day) plus aspirin (100 mg/day) or rabeprazole (20 mg/day) plus clopidogrel (75 mg/day) for 12 weeks. The primary end point is treatment success (ulcer healing rate). The secondary end point is incidence of ulcer bleeding within 12 weeks.

If rabeprazole plus aspirin in not inferior to rabeprazole plus clopidogrel in the incidence of ulcer healing and ulcer bleeding in the healing phase,PPI plus aspirin rather than PPI plus clopidogrel will be recommended during acute ulcer healing in patients who need antiplatelet therapy for their CV prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have taken aspirin for more than 1 month and are found to have PUD by upper endoscopy will receive PPI (rabeprazole 20 mg once daily) to treat their PUD. PUD in the upper gastrointestinal (UGI) tract is defined as

  * [1] mucosal break of stomach or duodenum > 3 mm in diameter; or
  * [2] more than 10 gastric or duodenal erosions, without malignancy proved by histopathological examination.

Exclusion Criteria:

* Patients will be excluded if they have PUD with bleeding (ulcer with adherent blood clot, visible vessel, oozing, or spurting) requiring endoscopic hemostasis,
* if they take other antithrombotic or anticoagulants simultaneously, if they have take NSAIDs, selective COX-2 inhibitors, or steroid,
* if they have take misoprostol or histamine receptor-2 antagonist (H2RA),
* if they have bleeding tendency (thrombocytopenia with platelet count < 80000/mm3 or prolonged pro thrombin time > 5 seconds),
* if they have anemia (hemoglobin < 10 g/dL),
* if they have received a surgical intervention due to PUD complication (bleeding, perforation, obstruction) in the past,
* if their age are > 80 year-old or < 18 year-old,
* if they have severe cardiovascular, pulmonary, hepatic, or renal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point is treatment success (ulcer healing rate). | 3 months

SECONDARY OUTCOMES:
The secondary end point is incidence of ulcer bleeding within 12 weeks. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Luo JC, Huang KW, Leu HB, Chen LC, Hou MC, Li CP, Lu CL, Lin HC, Lee FY, Lee SD. Randomised clinical trial: rabeprazole plus aspirin is not inferior to rabeprazole plus clopidogrel for the healing of aspirin-related peptic ulcer. Aliment Pharmacol Ther. 2011 Sep;34(5):519-25. doi: 10.1111/j.1365-2036.2011.04760.x. Epub 2011 Jul 5. PMID 21726257